CLINICAL TRIAL: NCT05392413
Title: Construction and Application of Immune Indicator Model for Predicting Efficacy of PD-1 Monoclonal Antibody in the Treatment of Advanced Esophageal Cancer
Brief Title: Immune Indicator Model for Predicting Efficacy of PD-1 Monoclonal Antibody
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-079
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Squamous Cell Carcinoma; PD-1 Inhibitor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- reactive group: According to the treatment effect, the patients were divided into two groups: reactive and non-reactive.
- non-reactive group: According to the treatment effect, the patients were divided into two groups: reactive and non-reactive.

SUMMARY:
200 patients with advanced esophageal cancer who received PD-1 monoclonal antibody treatment would be enrolled in this study. Changes in peripheral blood immune cells before and after treatment would be recorded and used for machine learning to establish a prediction model for the efficacy of PD-1 monoclonal antibody treatment.

DETAILED DESCRIPTION:
PD-1 monoclonal antibody has been used as a first-line drug for the treatment of advanced esophageal cancer, however, the ideal predictor of efficacy has not been established. The peripheral immune system plays an important role in driving anti-tumor effects, and the characteristics of peripheral immune cells can predict the effect of PD-1 monoclonal antibody therapy. However, the value of a single indicator for predicting the effect of PD-1 monoclonal antibody therapy is greatly limited. 200 patients with advanced esophageal cancer who received PD-1 monoclonal antibody treatment would be enrolled. Changes in peripheral blood immune cells before and after treatment would be recorded and used for machine learning to establish a prediction model for the efficacy of PD-1 monoclonal antibody treatment. The application between the indicator model and the expression level of PD-L1 in tumor tissue in predicting the efficacy of PD-1 monoclonal antibody in advanced esophageal cancer will be also study. This study aims to establish a peripheral blood immune cell-based models to predict the efficacy of PD-1 monoclonal antibody therapy for advanced esophageal cancer, provide a basis for guiding the selection of treatment options for advanced esophageal cancer, and improve the efficacy of PD-1 monoclonal antibody therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic advanced esophageal squamous cell carcinoma (stage IV) confirmed by histology or cytology who are ready to receive PD-1 monoclonal antibody combined with TP chemotherapy regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status score between 0 and 2.
* Have measurable lesions.
* Expected survival > 3 months.
* Subjects who have received anti-tumor therapy in the past should be enrolled after the toxicity of the previous treatment has returned to the baseline level (except for residual hair loss effects) or CTCAE v4.03 scale score ≤ 1.
* Female or male subjects of reproductive age and their partners should agree to use effective contraception from the time of signing the ICF until 6 months after the last dose of study drug.
* Absolute neutrophil count (ANC) ≥1.5×109/L, platelets ≥100×109/L, hemoglobin ≥9 g/dL. Liver: Bilirubin ≤1.5 times the upper limit of normal, alkaline phosphatase (AP) , Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 times the upper limit of normal (AP, AST, ALT ≤5 times the upper limit of normal are allowed if there is liver metastases) Renal: Calculated creatinine clearance ≥45 mL/min.

Exclusion Criteria:

* Have active, or have had an autoimmune disease that is likely to recur (eg, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, psoriasis, etc.) or at risk (e.g., organ transplant recipients requiring immunosuppressive therapy).
* Subjects who need to receive glucocorticoid (prednisone > 10 mg/day or equivalent dose of other similar drugs) or other immunosuppressive therapy due to certain conditions within 14 days prior to study drug administration.
* Major surgery, or radical radiation therapy, or palliative radiation therapy within the previous 14 days, or radiopharmaceuticals (strontium, samarium, etc.) within 56 days before starting study treatment.
* Received systemic anti-tumor therapy, including immunotherapy, biological therapy (tumor vaccines, cytokines, or growth factors to control cancer), etc. 14 days before starting study treatment.
* Have suffered from interstitial lung disease, chemical pneumonia, hypersensitivity pneumonitis, connective tissue disease pneumonia, pulmonary fibrosis, acute lung disease, etc. (except for local interstitial pneumonia induced by radiotherapy), or uncontrolled systemic disease, including diabetes and hypertension.
* Patients with human immunodeficiency virus (HIV) infection.
* patients with active pulmonary tuberculosis.
* Any active infection requiring systemic therapy by intravenous infusion within 2 weeks prior to the first dose of study drug.
* People who have received a solid organ transplant.
* Patients who have received any antibody/drug (including anti-programmed death-1 (PD-1), PD-L1, etc.) targeting T-cell co-regulatory proteins (immune checkpoints).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with advanced esophageal cell carcinoma who are ready to receive PD-1 monoclonal antibody therpy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
peripheral blood immune cells and immune molecules | 2022.1-2026.12
  Including absolute count of lymphocyte subsets, T lymphocyte subsets, B lymphocyte subsets, NK cell subsets, regulatory T cells, MDSC, etc. and IL-6, IL-10, etc.
Imaging examination | 2022.1-2026.12
  Including X-rays, CT, PET-CT and MR

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No